CLINICAL TRIAL: NCT05099484
Title: Medications in Breast Milk: A Convenience Pharmacokinetic Study (The MedMilk Study)
Brief Title: Medications in Breast Milk: A Convenience Pharmacokinetic Study
Acronym: MedMilk
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, Principle Investigator, Indiana University
Other Study IDs: 2001678776
Record Dates: First submitted 2021-10-05; First posted 2021-10-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from the participating mother and infant (if enrolled into study). Timing of collection will be dependent on the reported half-life of the DOI. Typically, 3 mL of blood will be obtained prior to dosing and at approximately 15, 30, 60, and 90 minutes, and 2, 4, 6, and 8 hours after taking the drug for most medications. If a woman is able to provide breast milk via a pump then approximately 3-15 mL of foremilk and hindmilk from each breast will be pumped at baseline (prior to dosing of drug) then at approximately 2, 4, 6, and 8 hours, or sooner if the subject experiences discomfort due to her breasts becoming engorged
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: The MedMilk study — This observational, pragmatic PK study will enroll lactating women who are taking medications that were prescribed by their treating medical provider or as an over-the-counter medication.

SUMMARY:
The benefits of breastfeeding and human milk consumption by infants has been clearly demonstrated. Benefits to the infant include reduction of infant and childhood diseases and allergies. Benefits to the woman include more rapid return to pre-pregnancy weight and reduced risk of health problems such as cardiovascular disease and diabetes in the future. Many women take medications as part of their standard of care and for multiple medical reasons in the postpartum period, when breastfeeding occurs. This creates a need for information about the transfer of drugs taken by a woman into breast milk, and ultimately, to the infant. Unfortunately, there are limited pharmacokinetic (PK) data on many of the medications commonly taken by lactating women. Additionally, there are little data on how the PK of drugs are impacted by lactation, and how this may vary from woman to woman or with time throughout lactation. Uptake of drugs into breast milk can vary due to a number of factors, including drug lipophilicity; molecular weight; drug half-life; active transport in breast epithelial cells; protein binding in milk and plasma; and lipid composition of breast milk. In silico and animal models can provide some information on transfer of drugs into breast milk, however, there are large gaps remaining in our knowledge of drug transfer into human milk. This information is crucial to better inform providers and patients about the transfer of those drugs to human breast milk. The purpose of this study is to characterize the PK of specific drugs of interest taken by lactating women as part of their standard of care. The drugs of interest (DOI) will be based on medical relevance and availability throughout the course of the study. The purpose of this study is to characterize the PK of medications taken by lactating women as part of their standard of care.

DETAILED DESCRIPTION:
This observational, pragmatic PK study will enroll lactating women who are taking medications that were prescribed by their treating medical provider or as an over-the-counter medication. Study investigators will not be prescribing or recommending medication use as part of this study. Feasibility of the study is enhanced by a partnership with The Milk Bank, which will refer women identified as taking medications to study investigators. Subjects will also be recruited from Eskenazi Health and IU Health. Blood and breast milk samples will be collected from lactating women prior to administration of a dose of drug and at varying time points after dosing to characterize maternal and infant plasma PK and transfer of drug into breast milk.

Another phase of the study will evaluate plasma concentrations of DOIs in breastfed infants whose mothers are already taking the medications. Infant blood samples will be obtained by heel stick or venipuncture from enrolled infants in order to determine the concentration of the drug in the infant's blood. The design of this study allows for the evaluation of the use of drugs in lactating women with minimal risk to participants. As blood draws and expressed milk samples are obtained often during clinical care or daily postpartum life, this study is not greater than minimal risk. Lactating women taking a DOI will have biospecimens collected from maternal breast milk and maternal blood. Breast milk will be collected from pumped or manually expressed samples.

ELIGIBILITY:
Inclusion Criteria:

* Women who are lactating, or who are admitted and/or consented for cesarean delivery and planning to breastfeed postpartum, AND are receiving at least one DOI per standard of care from their provider or through self-care (for over-the-counter medications).
* Mothers who are at least 18 years of age and no more than 45 years of age

Exclusion Criteria:

* Induced lactation
* Currently taking medication or supplements to increase milk production
* Diagnosis of any significant chronic medical condition including (but not limited to) hepatitis, HIV, heart failure, liver or renal failure, or malabsorption conditions (e.g. celiac disease or inflammatory bowel disease) known to alter PK of DOI, unless the DOI is the indicated treatment for that disease
* Alcohol use within 72 hours of study visit or planned PK blood draws
* Illicit substance, other than THC, use within 1 week of study visit or planned PK blood draws

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — breastfeeding female
Study Population: Approximately 50 lactating women and 50 infants receiving mother's breast milk will participate in this study. Approximately 20 to 50 eligible lactating women per DOI will be enrolled. Overall, the investigators intend to assay approximately 15-20 drugs. Participants may be enrolled for one or more DOIs with a single consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Drug concentration in maternal blood | study duration, typically up to 8 hours
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
Drug concentrations in breast milk at steady state | study duration, typically up to 8 hours
  Baseline and steady-state plasma concentrations of DOI in infants
Relative infant dose- drug concentration in infant blood sample | study duration, typically up to 8 hours
  calculation of relative infant dose

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, Principal Investigator — Indiana Univesity School of Medicine
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided